CLINICAL TRIAL: NCT00391651
Title: Short Course Nitrofurantoin For Acute Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Ann Stapleton, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20580-A; 01-1002-A 07
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Urinary Tract Infection
Keywords: UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Nitrofurantoin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nitrofurantoin 100mg BID x 5 days
  Interventions: Drug: Nitrofurantoin 100mg twice daily x 5 days; Drug: TMP/SMX DS twice daily x 3 days
- 2 (Active Comparator): TMP/SMX DS BID x 3 days
  Interventions: Drug: TMP/SMX DS twice daily x 3 days

INTERVENTIONS:
Drug: Nitrofurantoin 100mg twice daily x 5 days — Nitrofurantoin 100mg twice daily x 5 days
  Other Names: Macrobid
  Arms: 1
Drug: TMP/SMX DS twice daily x 3 days — TMP/SMX DS twice daily x 3 days
  Other Names: Septra

SUMMARY:
The purpose of this research study is to determine what the cure rates are with a 5 day course of nitrofurantoin versus the more standard 3 day course of trimethoprim/sulfamethoxazone. The study will improve our knowledge of which antibiotic and what length of therapy is best for treatment of UTI, taking into account the problem of antibiotic resistance.

Procedures subjects will undergo once they have read and signed the consent are:

Questions about their medical and sexual history and current symptoms of UTI. They will be asked to provide a urine sample and then randomly assigned to one of the two treatment groups.

will be obtained at each visit. If they were assigned to the nitrofurantoin treatment regimen, they will also be asked to collect a urine sample at home on the third day. If the subject develops recurrent urinary symptoms or does not have resolution of symptoms after completing the initial treatment course, they will be asked to return to the clinic and provide another urine sample for analysis. They will then be treated with another standard antibiotic at no cost to them and will be withdrawn from the study at that time.

The study population is women ages 18-45 with acute symptoms of a UTI without a history of UTI in the past 6 weeks.

DETAILED DESCRIPTION:
The purpose of this research study is to determine what the cure rates are with a 5 day course of nitrofurantoin versus the more standard 3 day course of trimethoprim/sulfamethoxazone. The study will improve our knowledge of which antibiotic and what length of therapy is best for treatment of UTI, taking into account the problem of antibiotic resistance.

Procedures subjects will undergo once they have read and signed the consent are:

Questions about their medical and sexual history and current symptoms of UTI. They will be asked to provide a urine sample and then randomly assigned to one of the two treatment groups. The randomization is generated by a Research Scientist working with the study.

They will be given a sheet to record symptoms at home. They will be asked to return to the clinic in 5-9 and 28-30 days after completing antibiotic therapy. Urine cultures will be obtained at each visit. If they were assigned to the nitrofurantoin treatment regimen, they will also be asked to collect a urine sample at home on the third day. If the subject develops recurrent urinary symptoms or does not have resolution of symptoms after completing the initial treatment course, they will be asked to return to the clinic and provide another urine sample for analysis. They will then be treated with another standard antibiotic at no cost to them and will be withdrawn from the study at that time.

The study population is women ages 18-45 with acute symptoms of a UTI without a history of UTI in the past 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years of age who were nonpregnant, in good general health, and had symptoms of acute cystitis (dysuria) and a urine culture with ³102 cfu/ml of a uropathogen

Exclusion Criteria:

* Women who were pregnant, lactating, or not regularly contracepting or with diabetes, had known anatomic abnormalities of the urinary tract, allergy to any of the study drugs, recent (<2 weeks) exposure to an oral or parenteral antimicrobial, or who were currently using prophylactic antibiotics were not eligible

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 338 (Actual)
Dates: Start 2002-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Microbiological Cure | 28-30 days post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Walter E Stamm, M.D., Principal Investigator — University of Washington; Kalpana Gupta, M.D., Principal Investigator — Yale University
Locations (1):
- University of WA, Seattle, Washington, United States

REFERENCES:
- [Result] Gupta K, Hooton TM, Roberts PL, Stamm WE. Short-course nitrofurantoin for the treatment of acute uncomplicated cystitis in women. Arch Intern Med. 2007 Nov 12;167(20):2207-12. doi: 10.1001/archinte.167.20.2207. PMID 17998493